CLINICAL TRIAL: NCT03093701
Title: TLC399 (ProDex) in Subjects With Macular Edema Due to Retinal Vein Occlusion (RVO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TLC399A2002
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Results first posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-11

CONDITIONS: Retinal Vein Occlusion; Macula Edema
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): TLC399 (ProDex) 0.36mg DSP with 100 mM PL
  Interventions: Drug: TLC399 (ProDex)
- Group 2 (Experimental): TLC399 (ProDex) 0.6 mg DSP with 100 mM PL
  Interventions: Drug: TLC399 (ProDex)
- Group 3 (Experimental): TLC399 (ProDex) 0.6 mg DSP with 50 mM PL
  Interventions: Drug: TLC399 (ProDex)
- Group 4 (Experimental): TLC399 (ProDex) 0.84 mg DSP with 50 mM PL
  Interventions: Drug: TLC399 (ProDex)

INTERVENTIONS:
Drug: TLC399 (ProDex) — 2-vial system: TLC399-DSP and TLC399-Lipid
  Other Names: TLC399

SUMMARY:
Randomized, double-masked trial designed to investigate the use of TLC399 (ProDex) in subjects with macular edema due to CRVO or BRVO.

DETAILED DESCRIPTION:
Part 1 is a randomized, double-maskedtrial trial designed to investigate the use of TLC399 in subjects with macular edema due to CRVO or BRVO. Three different dose strengths will be evaluated.

Part 2 is a randomized, double-masked study designed to evaluate 2 doses of TLC399 in subjects with macular edema due to CRVO or BRVO. Subjects will be randomized 1:1 to receive two different dose strenghs of investigational product.

ELIGIBILITY:
Inclusion Criteria:

1. male or female, at least 18 years of age
2. macular edema due to CRVO or BRVO
3. best-corrected visual acuity (BCVA) score of 20/40 to 20/400
4. mean central subfield thickness (CST) ≥350 um
5. willing and able to comply with the study procedure and sign a written informed consent
6. agree to use a medically acceptable form of birth control

Exclusion Criteria:

1. poorly controlled diabetes
2. history of significant intraocular pressure (IOP) elevation to steroid treatment
3. history of ocular hypertension and glaucoma
4. cataract surgery in the study eye within 3 months, or intraocular surgery within 6 months prior to screening
5. use of hemodilution for the treatment of RVO
6. use of IVT ranibizumab or bevacizumab in the study eye within 6 weeks prior to screening; or IVT aflibercept within 8 weeks prior to screening
7. IVT Ozurdex to the study eye within 6 months prior to screening
8. prior use of Retisert or Iluvien
9. use of systemic steroids or heparin within 1 month prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Shih, Study Director — Taiwan Liposome Company, Ltd.
Locations (20):
- United States (20):
  - Retinal Research Institute, Phoenix, Arizona
  - Retina Institute of California, Arcadia, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retina Institute of California, Palm Desert, California
  - Colorado Retina Associates, Golden, Colorado
  - Retina Group of New England, New London, Connecticut
  - Retina Macula Specialists of Miami, Miami, Florida
  - Georgia Retina, P.C, Marietta, Georgia
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Retina Consultants of Nevada, Las Vegas, Nevada
  - Retina Associates of Western New York, PC, Rochester, New York
  - Charlotte Eye Ear Nose & Throat Assoc, PA, Charlotte, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - Retina Research Institute of Texas, Abilene, Texas
  - Retina Research Center, Austin, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Retina Consultants of Houston,The Woodlands, The Woodlands, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 10 | 10 | 11 | 0
Completed | 10 | 7 | 11 | 0
Not Completed | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population was based on mITT population, which was defined as subjects who had at least 1 post-treatment efficacy evaluation
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 10 | 10 | 11 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (10.40) | 63.5 (12.55) | 68.5 (8.20) | 68.1 (10.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 1 | 8
  Male | 7 | 6 | 10 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 7
  Not Hispanic or Latino | 8 | 7 | 8 | 23
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 1 | 1 | 1 | 3
  White | 9 | 9 | 9 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 11 | 31
RVO Type [Count of Participants; unit: Participants]
  BRVO | 7 | 6 | 7 | 20
  CRVO | 3 | 4 | 4 | 11
CST (study eye) [Mean (Standard Deviation); unit: µm] | 530.6 (133.56) | 776.9 (288.67) | 702.1 (195.15) | 670.9 (231.75)
BCVA (study eye) [Mean (Standard Deviation); unit: letters] | 61.5 (7.40) | 48.2 (16.94) | 51.1 (16.66) | 53.5 (15.10)
IOP (study eye) [Mean (Standard Deviation); unit: mmHg] | 12.4 (2.63) | 13.5 (3.41) | 13.6 (2.69) | 13.2 (2.88)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With BCVA Gain of 15 or More Letters From Baseline in the Study Eye
Description: Proportion of subjects with BCVA gain of 15 or more letters from baseline in the study eye.
  Patients who received rescue medication/procedures within 6 months after the study treatment was initiated were considered failure to achieve a gain of at least 15 BCVA letters.
Time Frame: 6 months after dosing
Population: The analysis population was based on subject's randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 10 | 10 | 11
Participants | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: 14 days (screening) + 1 year
Description: Other (Not including serious) Adverse Events include both ocular (study eye only) and non-ocular adverse events.
  The safety population for AE reporting/analysis was based on the actual treatments received by the subjects.
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/8 | 1/13
Other Adverse Events (participants affected / at risk) | 10/10 | 8/8 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=10) | Group 2 (N=8) | Group 3 (N=13)
Vitreous haze (Eye disorders) | 0 | 1 | 0
Vitreous haze leading to significant vision loss (Eye disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Acute coliti (Gastrointestinal disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=10) | Group 2 (N=8) | Group 3 (N=13)
Vitreous haze (Eye disorders) | 10 | 8 | 13
Macular oedema (Eye disorders) | 4 | 2 | 5
Visual acuity reduced (Eye disorders) | 4 | 4 | 1
Conjunctival haemorrhage (Eye disorders) | 4 | 2 | 1
Vitreous floaters (Eye disorders) | 2 | 2 | 2
Vision blurred (Eye disorders) | 3 | 1 | 1
Corneal oedema (Eye disorders) | 1 | 1 | 1
Retinal vein occlusion (Eye disorders) | 0 | 0 | 2
Optic disc hyperaemia (Eye disorders) | 0 | 0 | 1
Retinal aneurysm (Eye disorders) | 1 | 0 | 1
Retinal vascular disorder (Eye disorders) | 0 | 1 | 1
Visual imparment (Eye disorders) | 1 | 0 | 1
Vitrous detachment (Eye disorders) | 0 | 2 | 0
Anterior chamber flare (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Cataract nulcear (Eye disorders) | 1 | 0 | 0
Conjunctival cyst (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Iris neovascularisation (Eye disorders) | 0 | 1 | 0
Macular fibrosis (Eye disorders) | 1 | 0 | 0
Macular pigmentation (Eye disorders) | 0 | 1 | 0
Maculopathy (Eye disorders) | 0 | 0 | 1
Retinal disorder (Eye disorders) | 1 | 0 | 0
Retinal exudates (Eye disorders) | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1
Retinal neovascularisation (Eye disorders) | 0 | 1 | 0
Retinal scar (Eye disorders) | 0 | 1 | 0
Vitreous disorder (Eye disorders) | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1
Vitreous opacities (Eye disorders) | 1 | 0 | 0
Retinal thickening (Eye disorders) | 1 | 1 | 0
Intraocular pressure increased (Investigations) | 2 | 3 | 4
Medication residue present (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 1
Cardiac murmur (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Heart rate irregular (Investigations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 3
Hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Glycosuria (Renal and urinary disorders) | 0 | 0 | 1
Nephropathy (Renal and urinary disorders) | 0 | 0 | 1
Renal artery occlusion (Renal and urinary disorders) | 0 | 0 | 1
Urine abnormality (Renal and urinary disorders) | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Dementia (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT03093701/Prot_SAP_000.pdf